CLINICAL TRIAL: NCT04835480
Title: A Phase II, Multicenter, Randomized, Positive-Controlled, and Multi-Cohort Study of OsrHSA in Patients With Decompensated Cirrhotic Ascites
Brief Title: A Phase II Study of OsrHSA in Patients With Decompensated Cirrhotic Ascites
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Healthgen Biotechnology Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: US-China-HY1001
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-04

CONDITIONS: Cirrhotic Ascites

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OsrHSA Group (Experimental): OsrHSA (10g or 20g), IV, qd
  Interventions: Drug: OrsHSA
- HSA Group1 (Active Comparator): HSA (10g or 20g), IV, qd
  Interventions: Drug: HSA

INTERVENTIONS:
Drug: OrsHSA — OsrHSA a recombinant HSA, which was expressed and purified from the plant Oryza sativa
  Arms: OsrHSA Group
Drug: HSA — Albutein® 20% (ALBUMIN HUMAN INFUSION 20% 50ML)
  Arms: HSA Group1

SUMMARY:
The study is designed to study the efficacy of IV OsrHSA or positive control HSA (10 g and 20 g IV everyday) for 14 days. After a screening period of up to 14 days, the eligible subjects will be randomized in a 4:1 ratio to OsrHSA and positive control HSA, respectively, in each cohort. Each enrolled subject will receive multiple assigned doses of OsrHSA. The Investigator and subjects will be blind to treatment assignment (OsrHSA or positive control HSA) in each cohort. During the study, subjects will be evaluated for efficacy, safety, tolerability, and immunogenicity. In each cohort, subjects will be stratified by baseline serum albumin level. If serum albumin reaches 35 g/L or more, the study drug or control drug administration may be terminated early. Subjects will have 3 follow-up visits in 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the ICF;
2. Decompensated cirrhosis with ascites by clinical, laboratory, or imaging evidence. Male or female eligible; Age ≥18 years and ≤80 years;
3. Serum albumin ≤30 g/L;
4. Has adequate venous access;
5. Be a female of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal and has a follicle stimulating hormone > 40mIU/mL, or surgically sterile [defined as having a bilateral oophorectomy, hysterectomy or tubal ligation]) or a woman of childbearing potential who agrees to one of the following to prevent pregnancy and has a negative serum pregnancy test at screening:

   * Practicing abstinence;
   * If a sexually active woman of childbearing potential (sexually active with a non-sterile male partner) agrees to prevent pregnancy by using double methods of contraception as follow until at least 90 days after the administration of the investigational product:

     * simultaneous use of the intrauterine contraceptive device, placed at least 4 weeks prior to study drug administration, and condom for the male partner;
     * simultaneous use of hormonal contraceptives, starting at least 4 weeks prior to study drug administration and must agree to use the same hormonal contraceptive throughout the study, and condom for the male partner;
     * simultaneous use of a diaphragm with intravaginally applied spermicide and male condoms for the male partner, starting at least 21 days prior to study drug administration.
   * Male subjects who are not vasectomized for at least 6 months and who are sexually active with a non-sterile female partner must agree to use double methods of contraception below from the first dose of randomized study drug until 90 days after their dose and must not donate sperm during their study participation period:

     * simultaneous use of a male condom and, for the female partner, hormonal contraceptives (used since at least 4 weeks) or intrauterine contraceptive device (placed since at least 4 weeks);
     * simultaneous use of a male condom and, for the female partner, a diaphragm with intravaginally applied spermicide.

Exclusion Criteria:

1. Previous known allergic/adverse reaction to cereal or any food containing cereal, including rice; A history of a severe allergic reaction to any HpHSA component or any food;
2. Positive IgE and IgG against rice at the screening, i.e. anti-rice Ig E ≥ 0.35 kU/L and anti-rice Ig G ≥ 25.0 mgA/L;
3. Subjects who have medical conditions except for hepatic cirrhosis, currently requiring the use of albumin such as paracentesis-induced circulatory dysfunction, large- volume paracentesis (>5 L each time);
4. Nephrotic syndrome, hepatorenal syndrome or Creatinine >2 × upper limit of normal (ULN), significant cardiopulmonary or structural heart disease, hemodialysis, active upper gastrointestinal bleeding, subjects with hepatic encephalopathy Grade III or IV (see Appendix 5 for hepatic encephalopathy stages);
5. Malignant ascites or ascites caused by cancer embolus;
6. Subjects with Grade C or D liver cancer according to the Barcelona-Clinic Liver Cancer staging (See Appendix 6);
7. Pregnancy;
8. HIV positive;
9. Active obstructive disease in the biliary tract defined by ultrasound or other imaging modalities;
10. With the following abnormal laboratory test values:

    Absolute neutrophil count (NE#) <1.0 × 109/L, platelets <30 × 109/L, white blood cells<2.0 × 109/L, hemoglobin <75 g/L; ALT and (or) AST >5 × ULN, total bilirubin > 5.0 ×ULN; PT INR > 2.0; Urine protein > 2+;
11. Subjects with Stage C or D heart failure according to ACCF/AHA Stage (See Appendix 7);
12. Previous transplant;
13. The mental state that prevents the subject from understanding the nature, extent, and consequences of the study;
14. Any clinical condition that the Investigator considers would make the subject unsuitable for the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
OrsHSA exhibits good efficacy by rescue serum albumin levels. | 14 days
  A relatively high percentage of subjects whose serum albumin reaches 35 g/L or more at any time up to 14 days by using OsrHSA.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Niu J, Gao Y, Wang G, Qin Z, Wu C, Yu Z, Wang L, Hu Z, Li X, Zhang Z, Chen Y, Yao L, Yang J, Li GM, Yang Y, Lu X, Gu Y, Wu X, Mao X, Zhou Z, Shang J, Lin B, Jia JD, Wang F, Zhang J, Ma H, Wang X, Yang CY, Yang D. Rice-derived recombinant human serum albumin as an alternative to human plasma for patients with decompensated liver cirrhosis: a randomised, double-blind, positive-controlled and non-inferiority trial. Gut. 2025 Aug 7;74(9):1476-1485. doi: 10.1136/gutjnl-2025-335577. PMID 40555465